CLINICAL TRIAL: NCT00045604
Title: A Phase I Study of Imatinib (Gleevec) in Combination With Irinotecan and Cisplatin in Extensive Stage Small Cell Lung Cancer
Brief Title: Imatinib Mesylate and Chemotherapy in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000256923; MSKCC-02015; NCI-5653
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2004-04

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Imatinib Mesylate; Irinotecan

INTERVENTIONS:
Drug: cisplatin
Drug: imatinib mesylate
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining imatinib mesylate with chemotherapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining imatinib mesylate with irinotecan and cisplatin in treating patients who have extensive-stage small cell lung cancer

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of imatinib mesylate when administered with irinotecan and cisplatin in patients with extensive stage small cell lung cancer.
* Determine the effect of imatinib mesylate on irinotecan metabolism by the cytochrome p450 system in these patients.
* Determine the response rate, time to progression, and survival of patients treated with this regimen.

OUTLINE: This is a dose-escalation study of imatinib mesylate.

Patients receive irinotecan IV over 30 minutes on days 1, 8, and 15 and cisplatin IV over 60 minutes on day 1. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients also receive oral imatinib mesylate once or twice daily beginning on day 22 of course 1 and continuing until disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of imatinib mesylate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 18 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed small cell lung cancer

  * Extensive stage disease
* Measurable or evaluable indicator lesion
* No symptomatic or uncontrolled brain or leptomeningeal involvement

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* WBC at least 4,000/mm3
* Platelet count at least 160,000/mm3
* Hemoglobin at least 10 g/dL

Hepatic

* Bilirubin no greater than 1 mg/dL
* AST no greater than 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 5 times ULN

Renal

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance at least 50 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No uncontrolled cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after study
* No other active cancer except previously treated carcinoma in situ, non -melanoma skin cancer, or stage I prostate cancer
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study
* No other concurrent uncontrolled illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy except for non-cancer conditions (e.g., low-dose methotrexate for rheumatoid arthritis)

Endocrine therapy

* Not specified

Radiotherapy

* At least 2 weeks since prior radiotherapy to major bone marrow-containing areas

Surgery

* Not specified

Other

* No concurrent warfarin for therapeutic anticoagulation

  * Low-molecular weight heparin or heparin allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-07

CONTACTS AND LOCATIONS:
Overall Officials: Lee M. Krug, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States